CLINICAL TRIAL: NCT06796491
Title: Effects of Post Isometric Relaxation and Post Facilitation Stretch on Pain, Range of Motion and Disability in Patients With Tight Hamstrings Syndrome
Brief Title: Effects of PIR and PFS on Pain, ROM, and Disabilty in Tight Hamstring Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0155
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hamstrings; Flexibility; Range of Motion; Disability
Keywords: Hamstrings; Flexibility; Muscle Energy Techniques; Range of motion; Post Facilitation Stretching; Post Isometric relaxation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Isometric Relaxation (Experimental): Patient applied the sub-maximal contraction almost 20%. Isometric contraction will be held for 10 seconds and then slight stretch for 30 seconds will be maintained. 4 contractions per treatment with 3 seconds rest between each contraction. This protocol continues 3 days/week for 4 weeks
  Interventions: Other: Post Isometric relaxation
- Post Facilitation Stretch (Active Comparator): Isometric contraction will be held for 10 seconds and then slight stretch for 30 seconds will be maintained. 4 contractions per treatment with 3 seconds rest between each contraction. This protocol continues 3 days/week 4 weeks. for hamstring flexibility
  Interventions: Other: Post Facilitation stretch

INTERVENTIONS:
Other: Post Isometric relaxation — Group A will receive Post Isometric Relaxation (PIR) Patient applied the sub-maximal contraction almost 20%. Isometric contraction was held for 10 seconds and then slight stretch for 30 seconds was maintained.4 contractions per treatment with 3 seconds rest between each contraction. This protocol continues 3 days/week for 4 weeks conventional treatment Hot pack for 10 minutes Pelvic bridging: The subjects will be asked to lie supine and with knee flexed and then raise the pelvis upward till the comfort then hold that position for 5 sec and repetitions were 10 times Cat and camel: The subjects will be requested to prone kneel and then take a deep breath from nose while making hump in the back (cat) and breathe out from mouth while curving the spine (camel) for 5 second 10 times repetitions
  Arms: Post Isometric Relaxation
Other: Post Facilitation stretch — Group B will receive Post Facilitation Stretch (PFS) Isometric contraction was held for 10 seconds and then slight stretch for 30 seconds was maintained. 4 contractions per treatment with 3 seconds rest between each contraction. This protocol continues 3 days/week 4 weeks. for hamstring flexibility conventional treatment Hot pack for 10 minutes Pelvic bridging: The subjects will be asked to lie supine and with knee flexed and then raise the pelvis upward till the comfort then hold that position for 5 sec and repetitions were 10 times Cat and camel: The subjects will be requested to prone kneel and then take a deep breath from nose while making hump in the back (cat) and breathe out from mouth while curving the spine (camel) for 5 second 10 times repetitions
  Arms: Post Facilitation Stretch

SUMMARY:
This randomized clinical trial aims to compare the effects of post-isometric relaxation (PIR) and post-facilitation stretch (PFS) on pain, range of motion, and disability in individuals with tight hamstring syndrome. Conducted at Riphah Rehabilitation Clinic, Lahore, participants aged 18-35 years with posterior thigh pain will be divided into two groups. Both groups will receive hot pack therapy and core strengthening exercises, with Group A receiving PIR and Group B receiving PFS. Outcomes will be assessed at baseline and after 4 weeks using NPRS, a disability questionnaire, and a goniometer, with data analyzed using SPSS version 25.

DETAILED DESCRIPTION:
Both PIR and PFS are subtypes of Muscle Energy Techniques (MET) that have shown potential in improving muscle flexibility and reducing discomfort. This study aims to address the impacts of PIR and PFS on pain, ROM, and disability in patients with tight hamstrings syndrome, providing valuable insights for clinical practice and enhancing the understanding of effective interventions for this common musculoskeletal issue.

The current literature on stretching techniques for musculoskeletal conditions reveals several gaps specifically relevant to the effects of Post Isometric Relaxation (PIR) and Post Facilitation Stretch (PFS) on tight hamstrings syndrome. Despite the high incidence of hamstring tightness and its association with conditions such as nonspecific low back pain, there is limited research directly comparing the effects of Post Isometric Relaxation (PIR) and Post Facilitation Stretch (PFS) on this condition. While studies have explored various stretching methods such as Muscle Energy Technique (MET), static stretching, and myofascial release, there is a notable lack of direct comparative research between PIR and PFS in patients with tight hamstrings. Additionally, existing studies had often focused on immediate or short-term outcomes, with limited investigation into the long-term effects of these techniques on pain, range of motion (ROM), and disability.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age between 18 to 35 years(45)
* Bilateral hamstring muscle tightness
* Individuals having lack of Active knee extension more than 20 degrees(46)

Exclusion Criteria:

* Low back pain radiating to the back of thigh
* History of fracture, dislocation of hip(47)
* Acute or chronic hamstring injury
* Any neurological disease(48)
* Congenital deformity of the lower limb
* Inflammatory condition that affects motion
* A history of a cervical whiplash injury(45)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-13 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4th week
  The severity of pain will be measured by using the NPRS scale, which goes from '0' (meaning there is no pain) to 10'' (meaning there is most agony possible) ("pain is severe as you can imagine"). It was accepted that the scale was convenient for determining patients' pain thresholds. The NPRS scale has a score range of 0 to 10. It was a valid and reliable tool. Va;idity ranging from 0.79 to 0.95 and reliability from 0.67 to 0.96.

SECONDARY OUTCOMES:
Active Knee Extension Test | 4th week
  AKE is an active test considered as a gold standard for hamstring flexibility assessment. The AKE test interrater reliability was excellent, with ICC2, values of 0.87 (0.58-0.97; 95%CI) for the dominant knee and 0.81 (0.41-0.94; 95%CI) for the nondominant knee and standard error of measurement (SEM) values of 3.5° (18.0°- 31.7°; 95%CI) and 3.8° (16.9°-31.7°; 95%CI) respectively. Minimal detectable change was between 9.7° and 10.5°. No significant difference in mean AKE measurements was noted between the first and second testing sessions for both raters (Table 4). The ICC3,1 values ranged from 0.78 to 0.92.
Modified Oswestry Disability Index | 4th week
  The Oswestry Disability Index (ODI) has become one of the principal condition-specific outcome measures used in the management of spinal disorders. The ODI remains a valid and vigorous measure of condition-specific disability. The authors recommend the use of version 2.0. The data presented are a guide to the power of the instrument to detect meaningful changes in disability status.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Shaukat, TDPT, Principal Investigator — Riphah International University
Locations (1):
- Zafar Hospital lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castellote-Caballero Y, Valenza MC, Puentedura EJ, Fernandez-de-Las-Penas C, Alburquerque-Sendin F. Immediate Effects of Neurodynamic Sliding versus Muscle Stretching on Hamstring Flexibility in Subjects with Short Hamstring Syndrome. J Sports Med (Hindawi Publ Corp). 2014;2014:127471. doi: 10.1155/2014/127471. Epub 2014 Apr 15. PMID 26464889
- [Background] Duhig S, Shield AJ, Opar D, Gabbett TJ, Ferguson C, Williams M. Effect of high-speed running on hamstring strain injury risk. Br J Sports Med. 2016 Dec;50(24):1536-1540. doi: 10.1136/bjsports-2015-095679. Epub 2016 Jun 10. PMID 27288515
- [Background] Woods C, Hawkins RD, Maltby S, Hulse M, Thomas A, Hodson A; Football Association Medical Research Programme. The Football Association Medical Research Programme: an audit of injuries in professional football--analysis of hamstring injuries. Br J Sports Med. 2004 Feb;38(1):36-41. doi: 10.1136/bjsm.2002.002352. PMID 14751943
- [Background] Rahnama N. Prevention of football injuries. Int J Prev Med. 2011 Jan;2(1):38-40. No abstract available. PMID 21448404
- [Background] Skoffer B. Low back pain in 15- to 16-year-old children in relation to school furniture and carrying of the school bag. Spine (Phila Pa 1976). 2007 Nov 15;32(24):E713-7. doi: 10.1097/BRS.0b013e31815a5a44. PMID 18007232
- [Background] Arab AM, Nourbakhsh MR. Hamstring muscle length and lumbar lordosis in subjects with different lifestyle and work setting: comparison between individuals with and without chronic low back pain. J Back Musculoskelet Rehabil. 2014;27(1):63-70. doi: 10.3233/BMR-130420. PMID 23948840
- [Background] Hollman JH, Berling TA, Crum EO, Miller KM, Simmons BT, Youdas JW. Do Verbal and Tactile Cueing Selectively Alter Gluteus Maximus and Hamstring Recruitment During a Supine Bridging Exercise in Active Females? A Randomized Controlled Trial. J Sport Rehabil. 2018 Mar 1;27(2):138-143. doi: 10.1123/jsr.2016-0130. Epub 2018 Mar 1. PMID 28121207
- [Background] Kumazaki T, Ehara Y, Sakai T. Anatomy and physiology of hamstring injury. Int J Sports Med. 2012 Dec;33(12):950-4. doi: 10.1055/s-0032-1311593. Epub 2012 Aug 15. PMID 22895873